CLINICAL TRIAL: NCT01025180
Title: Randomized Multicentre Prospective Study of Procalcitonin-guided Treatment on Antibiotic Use and Outcome in Severe Sepsis ICU Patients Without Obvious Infection
Brief Title: Study of Procalcitonin (PCT)-Guided Antibiotic Use in Severe Sepsis Patients Without Obvious Infection
Acronym: Pro-SEPS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 65 patients were included after 2 years instead of 140
Sponsor: Brahms France (Industry)
Responsible Party: Djillali Annane/ Professor, Coordinator and Principal Investigator
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PCT-F-2005-10
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2009-12

CONDITIONS: Severe Sepsis
Keywords: safety; Procalcitonin; PCT; SOFA; Sepsis; Antibiotic; Strategy; SIRS; severe sepsis without obvious infection
MeSH Terms: conditions — Sepsis | interventions — Procalcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procalcitonin level (Other): duration of the antibiotic treatment guided by procalcitonin level
  Interventions: Other: Procalcitonin level
- physician's appreciation (No Intervention): duration of the antibiotic treatment based on physician's appreciation

INTERVENTIONS:
Other: Procalcitonin level — The duration of antibiotic treatment is based on PCT level:
  * < 0.25 ng/ml: antibiotic should be stopped
  * 0.25 < PCT <0.5: antibiotic prescription is not recommended
  * > 0.5 ng/ml: antibiotic should be used
  Arms: Procalcitonin level

SUMMARY:
A recent study has demonstrated that in low respiratory infections, a strategy using prescription of antibiotics based on the pro-calcitonin level allows decreasing recourse to antibiotics by 47% without prognostic modification.

The aim is to evaluate the impact on antibiotics consumption of an algorithm using procalcitonin level in patients exhibiting severe sepsis symptomatology but without clearly identified hosted germs or infectious centre.

This multicenter study is a randomized prospective open study involving 9 ICU departments in France, comparing two strategies on antibiotherapy treatment period one based on procalcitonin level(experimental group) the other on physician's appreciation(control group)

140 adult patients should be included with a severe sepsis symptomatology, whose infectious etiology has not been proven. The main non-inclusion criterium is: the presence of a pathogen agent or infectious centre clearly identified.

The primary outcome is the rate of patients undergoing antibiotic treatment at D5.

Secondary outcomes: duration of the antibiotic treatment, mortality rate and duration in stay in intensive care ward and evolution of the SOFA score between D0, D3 and D5.

Duration of patient enrollment is 30 days.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in resuscitation ward
* severe sepsis symptomatology
* at least 2 SIRS criteria
* no infectious etiology detected
* at least one organ deficiency

Exclusion Criteria:

* the presence of a pathogen agent or infectious centre clearly identified
* pregnancy
* burned
* patients with therapeutic limitation
* recent surgery
* secondary neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
rate of patients undergoing antibiotic treatment at D5. | at D5

SECONDARY OUTCOMES:
evolution of the SOFA score between D0, D3 and D5. | D30

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, Professor, Principal Investigator — Raymond Poincaré hospital Garches-France
Locations (9):
- France (9):
  - ICU in J.Minjoz hospital, Besançon
  - ICU in Avicenne hospital, Bobigny
  - ICU in Ambroise Paré hospital, Boulogne
  - ICU in Raymond Poincaré hospital, Garches
  - ICU in André Boulloche hospital, Montbéliard
  - ICU in Centre hospitalier général, Mulhouse Belfort
  - ICU in St Etienne hospital, Saint-Etienne
  - ICU in Purpan hospital, Toulouse
  - ICU in Rangueil hospital, Toulouse